CLINICAL TRIAL: NCT04000464
Title: Comprehensive Lifestyle Improvement Program for Men With Prostate Cancer
Acronym: CLIPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1806697620
Record Dates: First submitted 2018-10-15; First posted 2019-06-27 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Pre and Post study model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): 24 Week Lifestyle Modification intervention
  Interventions: Behavioral: CLIPP

INTERVENTIONS:
Behavioral: CLIPP — Diabetes Prevention program and Comprehensive Lifestyle Improvement Program consisting of low calorie diet, physical activity, sleep optimization and stress management

SUMMARY:
This study is an investigator initiated clinical study. A prospective, single arm unblinded, open label study will be carried out to determine the feasibility of recruitment, retention and adherence of 30 prostate cancer survivors who have been on androgen deprivation therapy within the last 5 years for a lifestyle modification intervention.

DETAILED DESCRIPTION:
Introduction

* Androgen deprivation therapy (ADT) has been demonstrated to improve disease free and over-all survival in men with prostate cancer (PCa).
* ADT for PCa is associated with adverse cardio-metabolic effects such as reduced libido, hot flashes, metabolic syndrome, diabetes, myocardial infarction and stroke. This reduces quality of life (QoL) and potentially affects mortality.
* There is paucity of data regarding comprehensive lifestyle interventions in men on ADT for Pca. Existing studies used non-standardized interventions or lack data on metabolic risk factors.
* CLIPP is designed to address these gaps by using an intervention modelled after the Diabetes Prevention Program (DPP), a standardized multi-component intervention with demonstrated effectiveness in reducing diabetes risk factors that has been successfully adapted for multiple disease types including breast cancer.

Intervention:

* 24 Weeks
* Health Coaching Weekly
* Serum & Urine Baseline, Week 12 and Week 24
* Anthropometric Measures
* Questionnaires
* Dual-energy X-ray absorptiometry (DXA) at Baseline and Week 24

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with prostate cancer Stage I, II or IV
* On androgen deprivation therapy with last 5 years
* Willing to participate in a lifestyle modification program
* Willing to modify diet and eating practices
* Willing to participate in blood collection, urine collection and measurements
* Minimum of 30 days since participating in another study/trial
* English speaking
* 40 years of age or older

Exclusion Criteria:

* Currently participating in another study or trial
* Currently in hospice
* Inability to walk two city blocks
* Inability to comprehend informed consent or procedural requirements
* Digestive Diseases (IBD, Diverticulitis, etc) that might prevent him from increasing fruit and vegetable intake

Ages: 40 Years to 89 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Reach Recruiting Target | 6 Months
  Recruit 30 men with prostate cancer who have been on androgen deprivation therapy within the last 5 years.
Retention of Participants | 6 months
  80% retention rate, or 24 out of 30 participants
Adherence to Intervention | 6 months
  75% attendance rate throughout 24 intervention visits

SECONDARY OUTCOMES:
Fasting Glucose | 6 Months
  Unit of Measure Mg/dL
Lipid Panel | 6 Months
  Unit of Measure Mg/dL
Hemoglobin A1c | 6 Months
  Unit of Measure %
Global Quality of Life Questionnaire | 6 Months
  PROMIS Scale v 1.2 Global Health. Scale Measurements 1 to 5. 1=Poor 2=Fair 3=Good 4=Very Good 5= Excellent
Specific Quality of Life Questionnaire | 6 Months
  Expanded Prostate Cancer Index Composite Short Form (EPIC-26) - Scale of Measurement 0 to 4. 0=No Problem 1=Very Small problem 2=Small Problem 3=Moderate problem 4=Big Problem

OTHER OUTCOMES:
Inflammatory pathways associated with Prostate Cancer Progression. | 6 Months
  Inflammation markers measured will include Interleukin-6, Interleukin 1-beta, Interleukin-8, stromal cell derived factor 1-alpha & basic fibroblast growth factor.
Angiogenic pathways associated with prostate cancer progression | 6 Months
  Determine the effect of comprehensive lifestyle modification intervention on angiogenesis, markers, important mechanisms for prostate cancer progression using blood, serum and urine. Angiogenesis markers will include vascular endothelial growth factor & plasma placental growth factor) using Enzyme Linked Immunosorbent Assay (ELISA).

CONTACTS AND LOCATIONS:
Overall Officials: Amit Algotar, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona School of Medicine Collaboratory, Tucson, Arizona, United States